CLINICAL TRIAL: NCT04332861
Title: Evaluation of Infection in Obstructing Urolithiasis: A Prospective Observational Study
Brief Title: Evaluation of Infection in Obstructing Urolithiasis
Acronym: eIOU
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Margaret Pearle, Professor of Medicine, University of Texas Southwestern Medical Center
Other Study IDs: STU-2018-0028
Record Dates: First submitted 2020-03-30; First posted 2020-04-03 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Kidney Stone; Kidney Calculi; Urinary Tract Obstruction; Infection; Sepsis
Keywords: Kidney Stone; Kidney Calculi; Urinary Tract Obstruction; Infection; Sepsis
MeSH Terms: conditions — Kidney Calculi; Infections; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Excess/discarded blood specimens
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prospective observational cohort: For data analysis, the cohort will be subdivided as follows:
  * Identification and Validation cohorts
  * Patients with and without complicating factors
  * Patients with and without measured inflammatory marker levels
  Interventions: Other: Initial clinical and laboratory evaluation

INTERVENTIONS:
Other: Initial clinical and laboratory evaluation — Initial evaluation, prior to administration of any antibiotics if possible, includes history, physical exam, and labs including:
  * Urinalysis
  * Urine culture
  * Blood cultures
  * Complete blood count with differential
  * Comprehensive metabolic panel
  * Lactate
  * Procalcitonin
  * Other inflammatory markers

SUMMARY:
Obstructing urolithiasis can be life-threatening in the setting of urinary tract infection. The purpose of this study is to identify and validate risk factors and markers for the presence of infection and development of sepsis among patients with obstructing urolithiasis.

DETAILED DESCRIPTION:
An obstructing stone and suspected urinary tract infection is an indication for drainage of the renal collecting system. In this setting, decompression with a ureteral stent or percutaneous nephrostomy (PCN) is associated with decreased mortality and both methods have similar efficacy. At the time of initial evaluation, it is sometimes uncertain whether infection is present, resulting in difficult management decisions. It is also difficult to identify infected patients at greatest risk of developing sepsis, defined as life-threatening organ dysfunction caused by a dysregulated host response to infection.

There are currently no widely adopted criteria for the accurate diagnosis of infection in the setting of an obstructing stone. Abnormal vital signs, leukocytosis, and abnormal urinalysis are relied upon, but these findings are often indeterminate. Most studies to date addressing this problem have retrospectively evaluated associations of single variables with infection including pyuria and bacteriuria, or performance of sepsis screening tools such as the Sepsis-related Organ Failure Assessment (SOFA).

More accurate diagnostic measures for infected obstructing urolithiasis and a better understanding of its natural history are needed in order to improve patient outcomes. While early recognition of patients at significant risk of developing sepsis is essential, treatment of patients who are not clinically infected with antibiotics and decompression procedures is unnecessarily morbid. Therefore, the investigators aim to develop and validate diagnostic criteria to predict development of life-threatening infection in a prospective observational fashion.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18 and older
* Acute presentation of obstructing urolithiasis diagnosed on CT

Exclusion Criteria:

* Indwelling nephrostomy tubes or ureteral stents
* Staghorn calculi or evidence of xanthogranulomatous pyelonephritis

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects will be men and women presenting to the emergency department or already admitted to the hospital with a new diagnosis of obstructing urolithiasis on computed tomography (CT).
Sampling Method: Probability Sample
Enrollment: 477 (Actual)
Dates: Start 2019-09-03 (Actual); Primary Completion 2020-07-28 (Actual); Study Completion 2020-07-28 (Actual)

PRIMARY OUTCOMES:
Urinary tract infection (positive urine culture) | Within 24-72 hours of initial clinical and laboratory evaluation
  Urinary tract infection, defined as a positive urine culture
Intensive care unit admission and/or death due to sepsis during inpatient encounter | On average within 24-72 hours after initial clinical and laboratory evaluation
  Intensive care unit admission and/or death secondary to sepsis, occurring during the inpatient incounter.

SECONDARY OUTCOMES:
Bacteremia (at least one positive blood culture) | Within 24-72 hours of initial clinical and laboratory evaluation
  Bacteremia, defined as at least one positive blood culture
Pyonephrosis (drainage of pus from the involved kidney) during inpatient encounter | On average within 24-72 hours after initial clinical and laboratory evaluation
  Pyonephrosis, defined as drainage of pus from the involved kidney at any point during the inpatient encounter

CONTACTS AND LOCATIONS:
Overall Officials: Jodi Antonelli, MD, Principal Investigator — University of Texas Southwestern Medical Center; Margaret S Pearle, MD PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (2):
- United States (2):
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern Medical Center Clements University Hospital, Dallas, Texas

REFERENCES:
- [Background] Assimos D, Krambeck A, Miller NL, Monga M, Murad MH, Nelson CP, Pace KT, Pais VM Jr, Pearle MS, Preminger GM, Razvi H, Shah O, Matlaga BR. Surgical Management of Stones: American Urological Association/Endourological Society Guideline, PART I. J Urol. 2016 Oct;196(4):1153-60. doi: 10.1016/j.juro.2016.05.090. Epub 2016 May 27. PMID 27238616
- [Background] Borofsky MS, Walter D, Shah O, Goldfarb DS, Mues AC, Makarov DV. Surgical decompression is associated with decreased mortality in patients with sepsis and ureteral calculi. J Urol. 2013 Mar;189(3):946-51. doi: 10.1016/j.juro.2012.09.088. Epub 2012 Sep 24. PMID 23017519
- [Background] Pearle MS, Pierce HL, Miller GL, Summa JA, Mutz JM, Petty BA, Roehrborn CG, Kryger JV, Nakada SY. Optimal method of urgent decompression of the collecting system for obstruction and infection due to ureteral calculi. J Urol. 1998 Oct;160(4):1260-4. PMID 9751331
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] Abrahamian FM, Krishnadasan A, Mower WR, Moran GJ, Talan DA. Association of pyuria and clinical characteristics with the presence of urinary tract infection among patients with acute nephrolithiasis. Ann Emerg Med. 2013 Nov;62(5):526-533. doi: 10.1016/j.annemergmed.2013.06.006. Epub 2013 Jul 11. PMID 23850311
- [Background] Cheung F, Loeb CA, Croglio MP, Waltzer WC, Weissbart SJ. Bacteria on Urine Microscopy Is Not Associated with Systemic Infection in Patients with Obstructing Urolithiasis. J Endourol. 2017 Sep;31(9):942-945. doi: 10.1089/end.2017.0157. Epub 2017 Jun 27. PMID 28558478
- [Background] Fukushima H, Kobayashi M, Kawano K, Morimoto S. Performance of Quick Sequential (Sepsis Related) and Sequential (Sepsis Related) Organ Failure Assessment to Predict Mortality in Patients with Acute Pyelonephritis Associated with Upper Urinary Tract Calculi. J Urol. 2018 Jun;199(6):1526-1533. doi: 10.1016/j.juro.2017.12.052. Epub 2017 Dec 29. PMID 29291417